CLINICAL TRIAL: NCT04259671
Title: Exploring the Efficacy and Usability of the My Autism Passport (MAP) App in Service Navigation for Families of Children with Autism
Brief Title: Exploring the Efficacy and Usability of the My Autism Passport (MAP).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REB 18-168
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Families of children between 0-6 years of age with a new ASD diagnosis who have consented to the study will be randomly assigned to either the control group (standard of care) or the intervention group (provided the MAP app). They will be in their randomly assigned group for the entire duration of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given that MAP's use is to assist parents in communication and service navigation, clinicians will be informed by the study team which family has been allocated to the MAP group. For children allocated to the control group, clinicians will be instructed to continue with usual clinical care. In the Developmental Passport Pilot study, clinicians were blinded to the intervention and the study team found this was a limitation as families were not able to share aspects of their service navigation with their health care providers (Young et al, 2019). As such, we will not blind members of the clinical team to intervention but allow both the intervention and usual care to co-occur within the pragmatic, real life setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention- My Autism Passport App (Experimental): Families will be given the application to upload to their mobile device and will be provided information on how to use the App by the research team. The contact information for a member of the research team who will be able to provide technical support will be available on the consent form. Families will use the mobile application for a total of 18 months.
  Given that this is a pragmatic trial of a tool that tracks services, it also may be used to communicate service access to other providers.
  Interventions: Device: My Autism Passport (MAP) Application
- Control-Standard of care (No Intervention): Families in the control group will continue with standard of clinical care, and receive any of the usual supports their clinic and region provides, including access to physicians, service navigators, social workers, nurses, etc.

INTERVENTIONS:
Device: My Autism Passport (MAP) Application — Families will be given the application to upload to their mobile device and will be provided information on how to use the App by the research team. MAP is a mobile alternative to the paper version, and offers additional benefits such as the ability to set reminders, see regional developmental service agencies and other resources on a map, and directs the caregiver to information so that they may further their understanding about how to support their child.
  Arms: Intervention- My Autism Passport App

SUMMARY:
To address developmental service navigation by families of children with autism spectrum disorder (ASD) an innovative paper-based tracking tool called the Pediatric Developmental Passport (Passport) was created by Dr. Elizabeth Young at St. Michael's Hospital. The Passport was adapted through a partnership between St. Michael's hospital and Autism Films Inc. into a mobile application called My Autism Passport (MAP). MAP allows families to learn about, and manage publicly-funded ASD services from their mobile device. Users can locate resources within their region, and track their progress in accessing services across multiple service agencies. The user can also set reminders on MAP which will be synced with their calendars, record notes, and read short summaries of the services offered by regional agencies. In this way, the application keeps families engaged, and allows them to take control of their child's care.

The feasibility of the MAP mobile application will be assessed by clinicians and end users. Clinicians from five developmental diagnostic organizations that have more than one year of experience diagnosing and providing follow up care to children with ASD will be informed of the study and invited to participate in recruitment in their respective practices. Caregivers of a child that is given a new diagnosis of ASD will be invited to participate in the study and be randomized to the control group or non control group and may have access to the application for 18 months. During the 18 month period, data on how caregivers are using the app will be collected. At 6, 12 and 18 months, caregivers will be invited to participate in questionnaires on number of services accessed, parent stress levels and self-efficacy levels. Questionnaires and interviews will be quantitatively analyzed for differences between groups, and findings will be used to improve the app prior to a larger prospective clinical trial.

DETAILED DESCRIPTION:
Background: To improve service navigation, the investigators created a tool for caregivers to use to track their progress in accessing services called The Pediatric Developmental Passport (Passport). The Passport is a paper based tool that is modeled after the Ontario Immunization Record. It was developed using a mixed-methods Knowledge-to-Action framework that included participation from developmental pediatricians, pediatricians, and caregivers of children with ASD.

The Passport was pilot tested through a randomized control trial (RCT), at an academic health centre (academic), and a community clinic (community) Greater Toronto Area. Of the 40 families that received a new diagnosis of ASD, the proportion of families the contacted Applied Behaviour Analysis (ABA) services was 25% greater in the intervention (Passport) group than the placebo (dummy card) group. The contact rate for ABA services was also compared within each site. The academic site revealed no significant difference between the two groups. In the community site, 50% more families in the Passport group contacted ABA services when compared to the placebo group (p=0.019).Anecdotally, caregivers who had the Passport expressed appreciation and usability of the Passport as a tracking tool. In both the design and pilot phase of the study, caregivers identified that having the Passport available in an app form would facilitate its use, and enable them to use it more often and comprehensively.

Through a partnership with Autism Films the Passport has been developed into a mobile application called My Autism Passport (MAP). The development of this mobile Application was funded by the Telus Fund, TVO and the Manitoba Digital Media Tax Credit. MAP is a mobile alternative to the paper version, and offers additional benefits such as the ability to set reminders, see regional developmental service agencies and other resources on a map, and directs the caregiver to information so that they may further their understanding about how to support their child.

Similar to the Passport, the investigators now seek to evaluate the feasibility of MAP for use by caregivers in a real world setting. Given the success of the pilot RCT with the paper version of the Passport, the investigators seek to build on what the investigators learned through the pilot RCT using MAP. The results from this pilot RCT would be used to power a larger clinical trial.

Given the recent (April 2019) changes to Autism services, it is even more important to understand how families will navigate this new system for services. A control group would help inform prospectively how families will manage this new system of care, which may be different from how families managed in our previous Passport study. The intervention arm will help the investigators evaluate the effect of MAP in real time against this baseline.

Objectives of this pilot RCT are to evaluate if MAP: 1) increases the number of services families access over time and 2) decreases parental stress; 3) increases self-efficacy and 4) to provide data to inform sample size calculation for a full trial.

Methods Study Design A pragmatic, pilot randomized control trial will be conducted across 5 sites. The intervention will be use of MAP to help track services and the control group will receive standard of care including routine clinical follow ups.

Participant recruitment The study team will meet with clinicians, show them the intervention tool (MAP) and provide them with letters of information for their practices to hand out to eligible families. Alternatively, for practices identified as having a high volume of families with ASD, the research assistant (RA) will approach families in the waiting room identified by clinicians who may be eligible for the study. Interested families who meet inclusion criteria will be invited to participate in the study, will complete consent forms and initial demographic and parent stress and self-efficacy questionnaires.

Randomization Caregivers will be randomly assigned to the intervention or control group.

Intervention Families will be given the application to upload to their mobile device and will be provided information on how to use the App by the research team. Once consent has been obtained, participants will be provided with a study identification number which they will use to register for MAP.

Given that this is a pragmatic trial of a tool that tracks services, it also may be used to communicate service access to other providers. Therefore, caregivers will be able to discuss MAP and any other aspects of their follow up care with clinicians and other service providers. Clinicians will be informed by the RA as to which families have been given MAP to use.

Control Families in the control group will continue with standard of clinical care, and receive any of the usual supports their clinic and region provides, including access to physicians, service navigators, social workers, nurses, etc.

Data management A master-linking log matching families' last name and study ID will be kept in a double locked cabinet away separately from the data collection forms. The contact information for a member of the research team who will be able to provide technical support will be available on the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Families of children between 0-6 years of age, who have been diagnosed with autism spectrum disorder within the past month from five sites within the Greater Toronto Area that conduct developmental assessments will be eligible to participate in the study.

Exclusion Criteria:

* Caregivers who cannot read and communicate well enough in English to use an App.
* Caregivers who live outside of the greater toronto area.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Number of services contacted at 6 months | 6 months after diagnosis
  The number of services caregivers reported contacting
Number of services contacted at 12 months | 12 months after diagnosis
  The number of services caregivers reported contacting
Number of services contacted at 18 months | 18 months after diagnosis
  The number of services caregivers reported contacting

SECONDARY OUTCOMES:
Parental Stress Scale at 6 months | 6 months
  Caregivers will complete the Parent Stress Scale. This scale is a 18 item self report scale. Caregivers agree or disagree in terms of their typical relationship with their child or children on a 5 Point scale (strongly disagree, disagree, undecided, agree, strongly agree). The 8 positive items are reverse scored so that possible scores on the scale can range between 18-90. Higher scores indicate more stress (worse outcomes)
Parental Stress Scale at 12 months | 12 months
  Caregivers will complete the Parent Stress Scale. This scale is a 18 item self report scale. Caregivers agree or disagree in terms of their typical relationship with their child or children on a 5 Point scale (strongly disagree, disagree, undecided, agree, strongly agree). The 8 positive items are reverse scored so that possible scores on the scale can range between 18-90. Higher scores indicate more stress (worse outcomes)
Parental Stress Scale at 18 months | 18 months
  Caregivers will complete the Parent Stress Scale. This scale is a 18 item self report scale. Caregivers agree or disagree in terms of their typical relationship with their child or children on a 5 Point scale (strongly disagree, disagree, undecided, agree, strongly agree). The 8 positive items are reverse scored so that possible scores on the scale can range between 18-90. Higher scores indicate more stress (worse outcomes)
Parent Empowerment and Efficacy Measure at 6 months | 6 months
  Caregivers will complete the Parent Empowerment and Efficacy questionnaire. It is a 20 item list. The total possible score on this subscale ranges from 11 to 110 .The higher the score, the more positive the parent feels in their parenting role, in their personal growth as a parent and an individual, and in their achievement of goals shared by family. A higher score is a better outcome
Parent Empowerment and Efficacy Measure at 12 months | 12 months
  Caregivers will complete the Parent Empowerment and Efficacy questionnaire. It is a 20 item list. The total possible score on this subscale ranges from 11 to 110 .The higher the score, the more positive the parent feels in their parenting role, in their personal growth as a parent and an individual, and in their achievement of goals shared by family. A higher score is a better outcome
Parent Empowerment and Efficacy Measure at 18 months | 18 months
  Caregivers will complete the Parent Empowerment and Efficacy questionnaire. It is a 20 item list. The total possible score on this subscale ranges from 11 to 110 .The higher the score, the more positive the parent feels in their parenting role, in their personal growth as a parent and an individual, and in their achievement of goals shared by family. A higher score is a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Young, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, St.Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual research data will not be shared with other researchers.

REFERENCES:
- [Background] Young E, Aiyadurai R, Jegathesan T, Brown C, Bechard N, Minhas RS, Dillon K, Maguire J. Increasing Access to Developmental Services for Children with Autism Spectrum Disorder: The Pediatric Developmental Passport Pilot Randomized Trial. J Autism Dev Disord. 2019 Dec;49(12):4867-4876. doi: 10.1007/s10803-019-04199-3. PMID 31485815